CLINICAL TRIAL: NCT06550180
Title: The Additive Analgesic Effects of Transversus Abdominis Plane Block in Abdominoplasty Under Spinal Anaesthesia: A Randomized Controlled Study
Brief Title: The Additive Analgesic Effects of Transversus Abdominis Plane Block in Abdominoplasty Under Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, Principal Investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT2024-001
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-05

CONDITIONS: Abdominoplasty; Spinal Anaesthesia; Transversus Abdominis Plane Block (TAP Block)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal anaesthesia group (S) (Experimental): patient in S group They will receive 20 mg of 0.5% hyperbaric bupivacaine plus 25 microgram fentanyl.
  Interventions: Drug: Spinal anaesthesia group (S)
- oblique Subcostal TAP block and spinal anaesthesia group (OSTAP) (Experimental): Patients in (OSTAP) groups had spinal anesthesia administered with 20 mg of 0.5% hyperbaric bupivacaine and 25 mcg of fentanyl. Immediately after giving spinal anesthesia, individuals in the OSTAP group received 35 ml of 0.25% isobaric bupivacaine on each side.
  Interventions: Drug: Subcostal TAP block and spinal anesthesia group (STAP)

INTERVENTIONS:
Drug: Spinal anaesthesia group (S) — Spinal anaesthesia is given to all patients in S group. They will receive 20 mg of 0.5% hyperbaric bupivacaine plus 25 microgram fentanyl
  Arms: Spinal anaesthesia group (S)
Drug: Subcostal TAP block and spinal anesthesia group (STAP) — patient receive Subcostal TAP block before spinal anesthesia. Patients in STAP group will receive 20 ml of 0.25% isobaric bupivacaine for each side before spinal anesthesia
  Arms: oblique Subcostal TAP block and spinal anaesthesia group (OSTAP)

SUMMARY:
The primary outcome is the time to first request of opioid analgesia. The secondary outcomes are intraoperative analgesic needs, incidence of conversion to general anaesthesia, the total opioid dose in 24 hours, Visual analogue scale (VAS) scores at 2, 4, 6, 12, and 24 hours postoperatively, and the incidence of postoperative side effects (nausea, vomiting, hypotension, bradycardia, and pruritic).

DETAILED DESCRIPTION:
Abdominoplasty is designed to remove fat, skin laxity, and excess skin with the abdominal skin flap. It is a moderately invasive extraperitoneal procedure with or without liposuction. Ambulatory office-based abdominoplasty procedures have recently increased owing to lower cost and global availability of plastic surgeons in addition to better and safer anaesthetic techniques Spinal anaesthesia has many advantages such as pre-emptive analgesia, better control of pain, suppression of the surgical stress response, preservation of perioperative immune function, preservation of oxygenation and pulmonary functional residual capacity and improved visceral vascular flow in addition to reduction in the incidence of venous thrombotic disease and hence pulmonary embolism, as it facilitates early ambulation The addition of adjuvant drugs to local anesthetics and augmenting spinal anesthesia with peripheral nerve blocks would provide time for prolonged surgeries, and it is the ideal technique for procedures below T3-T4. The investigators assume that performing a transversus abdominis plane block (TAP block) just before spinal anesthesia in abdominoplasty would prolong the duration of postoperative analgesia and lessen the number of cases needing sedation or conversion to general anesthesia when compared to spinal anesthesia alone.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists physical status grade I and grade II.
* Age > 18 years and less than 65 years.
* Both sexes.

Exclusion Criteria:

* Patient refusal.

  -. Bleeding or coagulation abnormality.
* Local skin infection and sepsis at site of the block.
* Known hypersensitivity to the study drugs.
* Body Mass Index > 50 Kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the time to first request of opioid analgesia. | 24 hours
  assessment of pain by visual analogue scale (VAS) is a 10 cm horizontal line labeled "no pain" at one end and "worst pain" on the other end.

SECONDARY OUTCOMES:
total dose of intraoperative analgesic needs | 24 hours
  opioid dose by microgram

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian liver hospital, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.